CLINICAL TRIAL: NCT00258934
Title: Immunogenicity Study of the Influenza Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GID15
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Orthomyxoviridae Infections; Influenza
Keywords: Influenza; Orthomyxoviruses; Inactivated; Split-virion influenza vaccine; adults; Myxovirus Infection; Orthomyxovirus Infection
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Inactivated, split-virion influenza vaccine
- 2 (Active Comparator)
  Interventions: Biological: Inactivated, split-virion, influenza virus

INTERVENTIONS:
Biological: Inactivated, split-virion influenza vaccine — 0.1 mL single annual dose
  Arms: 1
Biological: Inactivated, split-virion, influenza virus — 0.5 mL single annual dose
  Other Names: Vaxigrip®
  Arms: 2

SUMMARY:
All marketed influenza vaccines are injected by the intramuscular (IM) route. This study will test whether an influenza vaccine is effective when injected by a route other than into the muscle. In order to prove this, the amount of antibodies in the blood will be measured before and after vaccination. In addition, the safety of both influenza vaccines will be tested by evaluating all serious reactions occurring after vaccination. The vaccine injected in this study is similar to the sponsor's marketed intramuscular influenza vaccine (Vaxigrip). In addition, the safety of both influenza vaccines administered by different routes will be tested by evaluating all adverse events and especially all serious reactions.

Primary Objective: To demonstrate and compare the immune response of an influenza vaccine after a single dose when administered by different routes.

Secondary Objectives: To describe the compliance of the immunogenicity of the vaccine with the European Medicine Agency (EMEA) after the first injection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 57 years on the day of inclusion
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative urine pregnancy test at V01
* For a woman of child-bearing potential: use of an effective method of contraception or abstinence for at least 4 weeks prior to, and at least four weeks after, the first vaccination.

At Year 1 (Visit 05):

-Addendum to the informed consent form signed and dated by the subject prior to vaccination at Visit 05

At Year 2 (Visit 07):

-Addendum to the informed consent form signed and dated by the subject prior to vaccination at Visit 07

Exclusion Criteria:

* Systemic hypersensitivity to egg proteins, chick proteins, or any of the vaccine components; in particular, neomycin, formaldehyde, and octoxinol 9, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Febrile illness (rectal equivalent temperature >= 38.0°C) on the day of inclusion
* Breast-feeding
* Participation in another clinical trial in the four weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency; immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months; or long-term systemic corticosteroid therapy.
* Chronic illness at a stage that could interfere with trial conduct or completion
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Blood or blood-derived products received in the past three months
* Any vaccination in the four weeks preceding the first trial vaccination
* Vaccination planned in the four weeks following the first trial vaccination
* Previous vaccination against influenza (in the previous six months) with the trial vaccine or another vaccine
* Thrombocytopenia or bleeding disorder contraindicating IM vaccination
* Subject deprived of freedom by an administrative or court order; or in an emergency setting; or hospitalized without his/her consent.

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 978 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of influenza vaccination. | 21 Days and 2 Years post-vaccination 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- Belgium (2):
  - Antwerp
  - Ghent
- Hamburg, Germany
- Allschwil, Switzerland

REFERENCES:
- [Derived] Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection (VAPI) questionnaire. Health Qual Life Outcomes. 2009 Mar 4;7:21. doi: 10.1186/1477-7525-7-21. PMID 19261173
- See also: Related Info — http://www.sanofipasteur.com